CLINICAL TRIAL: NCT01476891
Title: The eCALM Study - eTherapy for Cancer Applying Mindfulness: Online Mindfulness-Based Stress Reduction Program for Underserved Cancer Patients in Alberta: A Randomized Wait-list Controlled Trial.
Brief Title: The eCALM Study - An Online Mindfulness-Based Stress Reduction Program for Individuals Living With Cancer in Alberta
Acronym: eCALM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alberta Health services (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eCALM
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Mindfulness-Based Stress Reduction (MBSR); Cancer
Keywords: MBSR; Cancer; Online; Mindfulness Meditation; Randomized Waitlist Controlled Trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait-List (Active Comparator): Wait-list Control Group. The control group will receive the next available online MBSR program.
  Interventions: Other: Wait-list Control Group.
- Immediate MBSR (Active Comparator): Immediate Online MBSR Group. Participation in a standardized manual-based 8-week online MBSR program.
  Interventions: Other: Immediate MBSR

INTERVENTIONS:
Other: Immediate MBSR — Immediate Online MBSR Group. Participation in a standardized manual-based 8-week online MBSR program.
  Arms: Immediate MBSR
Other: Wait-list Control Group. — Wait-list Control Group. The control group will receive the next available online MBSR program.
  Arms: Wait-List

SUMMARY:
For people with cancer, in-person Mindfulness-Based Stress Reduction (MBSR) participation can decrease stress symptoms, mood disturbance, and fatigue, as well as enhance personal growth and spirituality, and improve quality of life and sleep. Online MBSR may improve the accessibility of MBSR programs to underserved cancer patients who are unable to attend available in-person groups. This study will examine whether patients are willing to participate and complete the program, and also whether the online program improves mood and stress.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak and read English sufficiently to complete questionnaires
* Women and men who have been diagnosed with any type of cancer, at any time in the past with no restriction on tumor site
* Pre or post primary cancer treatment, up to having completed primary cancer treatment within the last 36 months
* Exhibiting moderate distress
* Willing to participate in the intervention requirements; able to participate in the intervention (2 hrs per week for 8 weeks and a full day online retreat)
* Internet access
* Resident of Alberta, who has limited access to in-person cancer-specific MBSR programs

Exclusion Criteria:

* Presence of major self-reported psychiatric disorder not in remission, current substance abuse/dependence, and psychotic symptoms
* Previous participation in a MBSR program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 44 months
  recruitment, retention, attendance, adherence, satisfaction

SECONDARY OUTCOMES:
Efficacy | 44 months
  Profile of Mood States (POMS), Calgary Symptoms of Stress Inventory (C-SOSI)
Post-Traumatic Growth Inventory (PTGI) | 44 months
Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-Sp) | 44 months
Five Facet Mindfulness Questionnaire (FFMQ) | 44 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carlson, PhD, Principal Investigator — University of Calgary, Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Zernicke KA, Campbell TS, Speca M, McCabe-Ruff K, Flowers S, Carlson LE. A randomized wait-list controlled trial of feasibility and efficacy of an online mindfulness-based cancer recovery program: the eTherapy for cancer applying mindfulness trial. Psychosom Med. 2014 May;76(4):257-67. doi: 10.1097/PSY.0000000000000053. PMID 24804884
- [Derived] Zernicke KA, Campbell TS, Speca M, McCabe-Ruff K, Flowers S, Dirkse DA, Carlson LE. The eCALM Trial-eTherapy for cancer appLying mindfulness: online mindfulness-based cancer recovery program for underserved individuals living with cancer in Alberta: protocol development for a randomized wait-list controlled clinical trial. BMC Complement Altern Med. 2013 Feb 16;13:34. doi: 10.1186/1472-6882-13-34. PMID 23414206
- See also: Study Website — http://www.ecalm.ca
- See also: Investigator Website — http://www.lindacarlson.ca